CLINICAL TRIAL: NCT06051734
Title: Early Detection of Cardiac Affection in Patients of Wilson's Disease
Acronym: Wilson's
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salma Taha, Ass.Prof., Assiut University
Other Study IDs: Assiut University and Liver; Wilson's and heart (Registry Identifier: Wilson's and cardiac affection)
Record Dates: First submitted 2023-09-16; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Cardiovascular Diseases; Wilson's Disease
Keywords: Wilson's; CMR; Cardiac magnetic resonance
MeSH Terms: conditions — Cardiovascular Diseases; Hepatolenticular Degeneration

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Wilson disease (WD) is a rare autosomal recessive disorder caused by a genetic defect in ATP7B resulting in limited excretion of excess copper into the bile Pathological copper accumulation occurs in the entire body, with the liver and the brain being primarily affected

DETAILED DESCRIPTION:
Wilson disease (WD) is a rare autosomal recessive disorder caused by a genetic defect in ATP7B resulting in limited excretion of excess copper into the bile. Pathological copper accumulation occurs in the entire body, with the liver and the brain being primarily affected. The pathological copper accumulation may induce toxic injury, including mitochondrial dysfunction or apoptosis . Exhausted hepatic copper storage capacity causes copper release into the bloodstream thus affecting other organs, in particular the brain. The neurotoxicity of copper primarily damages astrocytes, leading to a regional destruction of the blood-brain barrier with subsequent neurological symptoms. Asymptomatic cardiac arrhythmias are quite common in WD. Cardiomyopathy, autonomic dysfunction, and cardiac deaths due to copper accumulation in cardiac tissue have occasionally been reported in WD. Copper accumulation induces toxic effects in cardiomyocytes and the clinical consequences of these myocardial accumulations are poorly understood. Previous studies have mainly reported mild cardiac abnormalities including concentric hypertrophy, impaired left ventricular (LV) relaxation and minor electrocardiographic changes, mainly reported in the times before appropriate treatment was available. A longitudinal cohort study demonstrated a higher incidence of heart failure (HF) and atrial fibrillation in WD patients, indicating a potential adverse effect of copper on the heart. Cardiovascular magnetic resonance (CMR) allows for a non-invasive tissue characterization, specifically visualizing edema, fibrosis, and pathological infiltrations. CMR has been successfully used for diagnosis and therapy monitoring in other storage diseases such as myocardial iron overload and amyloidosis. Survival in patients with thalassemia major improved significantly after the introduction of CMR for identifying myocardial iron accumulation. Imaging regional fibrosis using CMR late gadolinium enhancement (LGE) and quantitative measurement of extracellular volume (ECV) provide independent prognostic markers in cardiac amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with Wilson's

Exclusion Criteria:

* Claustrophobia
* Refusal to share information
* Heart failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with Wilson's disease attending outpatient clinic
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
evaluate spectrum of cardiac affection by copper deposition in Wilson disease patients and detect early cardiac affection | 1 year
  Evaluate the effect of copper on EF and diastolic function of LV and RV

IPD SHARING:
Plan to Share IPD: Undecided